CLINICAL TRIAL: NCT02254603
Title: To Evaluate the Effects of Weight-loss by the Combined Therapy of Acupuncture and Yoga Exercise
Brief Title: The Effects of the Combined Therapy of Acupuncture and Yoga Exercise on Weight Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Bing Show Chwan Memorial Hospital (Other)
Responsible Party: Principal Investigator, Shu-Hui Yeh, RN, PhD, Professor, Chang Bing Show Chwan Memorial Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1011003
Record Dates: First submitted 2014-09-25; First posted 2014-10-02 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-09

CONDITIONS: Obesity
Keywords: Obesity, ayuveda yoga exercise, acupuncture.
MeSH Terms: conditions — Obesity | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture controls (Other): Acupuncture group will receive 30-minutes treatment three times a week for 3 months.
  Interventions: Device: Acupuncture
- acupuncture and yoga exercise (Experimental): Subject will receive a combination of acupuncture and yoga exercise three times a week for 3 months.
  Interventions: Device: Acupuncture; Behavioral: Yoga exercise

INTERVENTIONS:
Device: Acupuncture — Acupuncture about 30 mins will be performed by a traditional Chinese physician three times a week for 3 months.
Behavioral: Yoga exercise — Subject will receive regular 60-minutes yoga exercise three times a week for 3 months.
  Arms: acupuncture and yoga exercise

SUMMARY:
The aim of this study is to examine the effects of combination of acupuncture and ayuveda yoga exercise on weight loss for the overweight.

DETAILED DESCRIPTION:
Obesity is a common health problem in developed countries. At present,the medical staff have already been alerted that the obesity is a kind of disease actually and one of the epidemic diseases which erode the human health in the world. It is not only about the person's health but also a main public health problem. It has been caught to our attention that some diseases, such as cardiovascular diseases,diabetes, and high blood pressure are coming along with overweight and obesity. Recent studies had demonstrated a positive correlation between chronic diseases and obesity. There are many treatments for the obesity, in general, acupuncture may be an effective one. Acupuncture may suppress the people's appetite, slow down the stomach's creeping motion, and increase the stomach's evacuation time. Simultaneously, acupuncture controls the body through the absorption and storage of the calorie via the adjustment of the endocrine system. But we still need a more efficiency way to accelerate the body fat metabolism and decrease the storage of the fat in vivo. Therefore, the purpose of this study is to examine the effects of combination of acupuncture and ayuveda yoga exercise on weight loss among the overweight.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 24

Exclusion Criteria:

* Diagnosis of cancer.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Reduce body mass index. | Change from baseline in body mass index at 3 months
  Outcome measure compares the change in body mass index during 3 months treatment.

SECONDARY OUTCOMES:
Reduce waistline | Change from baseline in waistline at 3 months
  Outcome measure compares the change in waistline during 3 months treatment.
Change biochemical profile of blood | Change from baseline in biochemical profile of blood at 3 months
  Outcome measure compares the changes in biochemical profile of blood including cholesterol/high-density lipoprotein/low-density lipoprotein/blood sugar during 3 months treatment. Peripheral blood will be collected at 2 different times. (1) baseline data: before intervention, (2) outcome data: at 3 months post-intervention.
Immune modulation | Change from baseline in lymphocyte profile and polarization at 3 months
  Immune function will be assessed by blood analysis including lymphocyte subpopulations (Th1/ Th2/ Treg/ Th17), polarization (T-bet/ Gata-3/ Foxp3/ RORrt), its related cytokines (Th1: IL-12/ IFN-γ/ IL-27; Th2: IL-4/ IL-13/ IL-25; Th17: IL-17A/ IL-6/ IL-21; Treg: TGF-β/ IL-10) during 3 months treatment. Peripheral blood will be collected at 2 different times. (1) baseline data: before intervention, (2) outcome data: at 3 months post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Kuender D. Yang, PhD., Study Chair — Chang Bing Show Chwan Memorial Hospital; Shu-Hui Yeh, PhD., Study Director — Chang Bing Show Chwan Memorial Hospital & Central Taiwan University of Science and Technology; Yu-Kwan Lu, MD., Principal Investigator — Show Chwan Memorial Hospital
Locations (1):
- Division of Core Laboratory; Chang Bing Show Chwan Memorial Hospital, Changhua County, Taiwan